CLINICAL TRIAL: NCT04055636
Title: Prospective Multidisciplinary Observational Trial of Cardiotoxicity in Patients Undergoing Anticancer Therapy.
Brief Title: Observational Trial of Cardiotoxicity in Patients Undergoing Chemotherapy.
Acronym: PROMETEY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Sponsor
Other Study IDs: PR_01
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-09

CONDITIONS: Cardiotoxicity; Heart Failure; Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiotoxicity; Heart Failure; Cardiomyopathy, Dilated | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, plasma.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- cancer survivors with heart failure and/or fatal arrhythmias: Patients undergoing cancer therapy for the last 3-4 years with signs of heart failure and/or life-threatening arrhythmias. Administered interventions: physical examination, echocardiography with speckle tracking analysis, 48-hour ECG monitoring, blood samples analysis for biochemistry, biomarkers of myocardial damage, fibrosis and inflammation.
  Interventions: Diagnostic Test: Echocardiography with speckle tracking analysis.; Diagnostic Test: 48-hour ECG monitoring.; Diagnostic Test: Blood samples analysis.
- Cancer survivors without complications: Patients undergoing cancer therapy for the last 3-4 years without signs of heart failure and/or life-threatening arrhythmias. Administered interventions: physical examination, echocardiography with speckle tracking analysis, 48-hour ECG monitoring, blood samples analysis for biochemistry, biomarkers of myocardial damage, fibrosis and inflammation.
  Interventions: Diagnostic Test: Echocardiography with speckle tracking analysis.; Diagnostic Test: 48-hour ECG monitoring.; Diagnostic Test: Blood samples analysis.
- Cancer patients before chemotherapy: Cancer patients before administered chemotherapy. Interventions: physical examination, echocardiography with speckle tracking analysis, 48-hour ECG monitoring, blood samples analysis for biochemistry, biomarkers of myocardial damage, fibrosis and inflammation.
  Interventions: Diagnostic Test: Echocardiography with speckle tracking analysis.; Diagnostic Test: 48-hour ECG monitoring.; Diagnostic Test: Blood samples analysis.
- Patients with non-toxic dilated cardiomyopathy (control).: Patients with non-toxic dilated cardiomyopathy. Administered interventions: physical examination, echocardiography with speckle tracking analysis, 48-hour ECG monitoring, blood samples analysis for biochemistry, biomarkers of myocardial damage, fibrosis and inflammation.
  Interventions: Diagnostic Test: Echocardiography with speckle tracking analysis.; Diagnostic Test: 48-hour ECG monitoring.; Diagnostic Test: Blood samples analysis.

INTERVENTIONS:
Diagnostic Test: Echocardiography with speckle tracking analysis. — Transthoracic echocardiography with speckle tracking analysis.
Diagnostic Test: 48-hour ECG monitoring. — Ambulatory 48-hour electrocardiography monitoring.
Diagnostic Test: Blood samples analysis. — Analysis of blood samples for biochemistry, biomarkers of myocardial damage, fibrosis and inflammation.

SUMMARY:
Advances in treatment have led to improved survival of patients with cancer, but have also increased morbidity and mortality due to cancer treatment side effects. Cardiotoxicity is one the most frequent side effect which may lead to premature morbidity and death among cancer survivors. The most concerning cardiovascular complications of cancer therapy is myocardial dysfunction, leading to heart failure, and fatal arrhythmias, especially those induced by QT-prolonging drugs.

PROMETEY (PROspective Multidisciplinary obsErvational Trial of cardiotoxicity in patiEnts undergoing anticancer therapy) - is Russian multicenter observational study assessing cardiotoxicity and its clinical, biochemical and genetic factors in patients on cancer therapy.

The objectives of the study are:

* to reveal prevalence of cardiotoxic effects of cancer therapy in routine clinical practice in Russian Federation,
* to assess contribution of these effects to mortality of patients on cancer therapy,
* to evaluate clinical and economic consequences of cardiotoxicity in patients with cancer,
* to develop an individualized model of cardiotoxicity risk factors based on clinical and laboratory parameters.

Patients: 400 cancer patients with toxic cardiomyopathy and 100 patients with idiopathic or family dilated cardiomyopathy.

Study duration: 60 months. All patients will undergo complex examination after signing informed consent form(ICF): physical exam, echocardiography with speckle tracking analysis, ambulatory 48-hours ECG monitoring, biochemistry, analysis of biomarkers of myocardial injury, fibrosis and inflammation.

Primary endpoint: all-cause mortality, heart transplantation, cardioverter-defibrillator implantation, hospitalization with heart failure decompensation.

Secondary endpoints:

* thromboembolism,
* fatal/ nonfatal myocardial infarction, stroke,
* sudden cardiac death,
* surgical therapy of heart failure or arrhythmias,
* cardiovascular death,
* all-cause mortality,
* heart transplantation,
* cardioverter-defibrillator implantation.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent form (ICF),
* Eastern Cooperative Oncology Group (ECOG) scale 0-3,
* patients with verified cancer on or planned to be on chemotherapy including anthracyclines,
* sufficient bone marrow function, including: absolute neutrophils > 1.5*10^9/l, platelets > 100*10^9/l, hemoglobin > 9 g/dl,
* sufficient liver function, including: total bilirubin < 1.5*upper normal value, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 upper normal value,
* sufficient renal function, including: creatinine clearance > 50 ml/min.

For control group:

* verified non-toxic dilated cardiomyopathy.

Exclusion Criteria:

* refusal of patient,
* sepsis,
* coma, delirium,
* mental disorders,
* left chest radiation therapy,
* metastases in central nervous system.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female more than 18 years old with verified cancer or with non-toxic dilated cardiomyopathy (control group).
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-06-14 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | During all observational period (60 months)
  Death of patient from all causes.
Heart transplantation | During all observational period (60 months).
  Heart transplantation associated with heart failure or toxic cardiomyopathy decompensation.
Cardioverter-defibrillator implantation | During all observational period (60 months).
  Implantation of cardioverter-defibrillator associated with life-threatening ventricular arrhythmias.
Hospitalization with heart failure decompensation | During all observational period (60 months)
  Hospitalization of patient due to decompensation of heart failure.

SECONDARY OUTCOMES:
Thromboembolism. | During all observational period (60 months).
  Venous thromboembolism associated with cancer disease.
Myocardial infarction | During all observational period (60 months).
  Fatal/nonfatal myocardial infarction.
Stroke | During all observational period (60 months).
  Stroke
Sudden cardiac death | During all observational period (60 months).
  Sudden cardiac death associated with fatal arrhythmias.
Surgical therapy of heart failure or arrhythmias | During all observational period (60 months).
  Surgical therapy of heart failure or arrhythmias.
Cardiovascular death | During all observational period (60 months).
  Death of patient associated with cardiovascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: Yury A Vasyuk, MD, Principal Investigator — Moscow State University of Medicine and Dentistry
Locations (1):
- Moscow State University of Medicine and Dentistry, Department of Hospital Therapy №1, Moscow, Moscow Oblast, Russia

IPD SHARING:
Plan to Share IPD: No